CLINICAL TRIAL: NCT04311736
Title: Concurrent Aerobic Exercise and Cognitive Training to Prevent Alzheimer's in At-risk Older Adults (The Exergame Study)
Brief Title: Concurrent Aerobic Exercise and Cognitive Training to Prevent Alzheimer's in At-risk Older Adults
Acronym: Exergames
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moai Technologies LLC (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EXERGAMES2
Record Dates: First submitted 2019-10-17; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Mild Cognitive Impairment; Exercise Training
Keywords: mild cognitive impairment; cognitive decline; aerobic exercise; physical exercise; exercise training; cognitive exercise; cognitive games; virtual reality
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergame (Active Comparator): Moderate intensity cycling only 3 times per week for 12 weeks + concurrent virtual reality cognitive training, supervised by an exercise specialist
  Interventions: Behavioral: Exergame
- Cycling (Active Comparator): Moderate intensity cycling only 3 times per week for 12 weeks, supervised by an exercise specialist
  Interventions: Behavioral: Cycling
- Stretching (Sham Comparator): Stretching 3 times per week for 12 weeks, supervised by a therapist
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Exergame — Cycling on a recumbent cycle ergometer + Virtual Reality Cognitive Training
  Arms: Exergame
Behavioral: Cycling — Cycling on a recumbent cycle ergometer
  Arms: Cycling
Behavioral: Stretching — Stretching exercises
  Arms: Stretching

SUMMARY:
In this research, a unique "Exergame" has been developed and is being tested. The Exergame consists of unique Virtual Reality Cognitive Training (VRCT) games combined with concurrent cycling on a recumbent stationary cycle. The Exergame seamlessly integrates specific cognitive tasks into a virtual environment and is synchronized with cycling to promote cognition. Cycling through an interesting virtual environment will motivate and engage the older adult to participate in the exercise, and VRCT could augment cycling's effects on cognition. A further innovation is that the Exergame has been developed as both an Apple TV and iPAD application, making it widely accessible and available. It will provide a low-cost VRCT Exergame option that currently does not exist, one that is affordable and compatible with almost any stationary cycle. This project is significant because treatment that delays the onset of Alzheimer's Disease (AD) by five years could save the U.S. economy an estimated $89 billion by 2030 and no drugs can yet prevent, cure, or even slow AD. Aerobic exercise and cognitive training are two such promising interventions. Emerging mechanistic studies further suggest that the two interventions together may have a synergistic, superior cognitive effect than either intervention alone. The purpose of this project is to demonstrate the feasibility and efficacy of the Exergame intervention on cognition. An RCT is planned in which subjects are randomized on a 2:1:1 allocation ratio to 3 parallel groups (exergame:cycling only:attention control). Mixed methods will be used to assess outcomes in both phases.

DETAILED DESCRIPTION:
A treatment that delays the onset of Alzheimer's disease (AD) by five years could be hugely cost-saving at an estimated $89 billion in 2030. However, nearly all (99.6%) drug trials for AD have failed, and no drugs can yet prevent, cure, or even slow AD. This highlights an urgent and pressing need to develop behavioral interventions to prevent AD and slow its progression. Aerobic exercise and cognitive training are two such promising interventions.

Aerobic exercise and cognitive training are 2 promising interventions for preventing AD. Aerobic exercise increases aerobic fitness, which in turn improves brain structure and function, while cognitive training improves selective neural function intensively. Hence, concurrent aerobic exercise and cognitive training may very well have an additive or synergistic effect on cognition by complementary strengthening of different neural functions because aerobic exercise and virtual reality cognitive training depend on discrete neuronal mechanisms for their therapeutic effects.

The purpose of this Phase II randomized controlled trial (RCT) is to test the efficacy and additive/synergistic effects of a 3-month combined cycling and virtual reality cognitive training intervention on cognition and relevant mechanisms (aerobic fitness, physical function), in persons with subjective cognitive decline at risk for developing AD.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive complaint (defines as answering yes to the question "Do you feel that your memory or thinking skills have gotten worse recently within the last 2 years?");
2. Not engaging in aerobic exercise or cognitive training >2 days/week, 30 minutes a session in the past 3 months;
3. Age 65 years and older;
4. Written consent.
5. Medical clearance to participate in a supervised exercise program

Exclusion Criteria:

1. Resting heart rate > 100 or <50 beats/min with symptoms;
2. Dementia or mild cognitive impairment (self-report, diagnosis, or scoring <26 on the Telephone Interview for Cognitive Status;
3. Evidence that cognitive decline or memory complaints were caused by underlying neurological or psychiatric disorder or chemical dependency as determined by primary health care provider;
4. Current enrollment in another intervention study;
5. ACSM contraindications to exercise or other factors that make exercise impossible or unsafe.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Episodic Memory | change from baseline to 3 months
  change in composite scores of episodic memory. Score are automatically computed by NIH Toolbox App,Scoring Process: Item Response Theory (IRT) is used to score the TPVT. A score known as a theta score is calculated for each participant; it represents the relative overall ability or performance of the participant. A theta score is very similar to a z-score, which is a statistic with a mean of zero and a standard deviation of one.

SECONDARY OUTCOMES:
Executive Function | change from baseline to 3 months
  change in composite measures of executive function, Score are automatically computed by NIH Toolbox App,Scoring Process: Item Response Theory (IRT) is used to score the TPVT. A score known as a theta score is calculated for each participant; it represents the relative overall ability or performance of the participant. A theta score is very similar to a z-score, which is a statistic with a mean of zero and a standard deviation of one.
Global Cognition | change from baseline to 3 months
  change in composite measures of global cognition. Score are automatically computed by NIH Toolbox App,Scoring Process: Item Response Theory (IRT) is used to score the TPVT. A score known as a theta score is calculated for each participant; it represents the relative overall ability or performance of the participant. A theta score is very similar to a z-score, which is a statistic with a mean of zero and a standard deviation of one.
Aerobic Fitness | change from baseline to 3 months
  change in 10 meter shuttle walk test

OTHER OUTCOMES:
Physical Function | change from baseline to 3 months
  change in 6 minute walk test
Physical Function | change from baseline to 3 month
  change in Short Physical Performance Battery Score-Balance
Physical Function | change from baseline to 3 months
  change in short physical performance battery score-Sit to stand
Physical Function | change from baseline to 3 months
  change in short physical performance battery score-4 meter Gait speed

CONTACTS AND LOCATIONS:
Overall Officials: Dereck L Salisbury, PhD, Principal Investigator — salis048@umn.edu
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salisbury DL, Pituch KA, Yu F. The Effects of Exergame Telerehabilitation in Persons With Subjective Cognitive Decline. Gerontologist. 2024 Jun 1;64(6):gnae028. doi: 10.1093/geront/gnae028. PMID 38486359
- [Derived] Salisbury D, Plocher T, Yu F. Efficacy of simultaneous aerobic exercise and cognitive training in subjective cognitive decline: study protocol for randomized controlled trial of the Exergames Study. Trials. 2021 Jan 6;22(1):14. doi: 10.1186/s13063-020-04950-7. PMID 33407727